CLINICAL TRIAL: NCT03036917
Title: Cognitive Function Before and After Opioid Reduction in Patients With Chronic Pain A Prospective Cohort Study
Brief Title: Cognitive Function Before and After Opioid Reduction in Patients With Chronic Pain
Acronym: coffee-cup
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SE-4-2016
Record Dates: First submitted 2017-01-10; First posted 2017-01-31 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2018-07

CONDITIONS: Chronic Nonmalignant Pain; Cognitive Impairment; Opiate Dependence
MeSH Terms: conditions — Cognitive Dysfunction; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to investigate the cognitive function of patients in the opioid reduction programme at the multidisciplinary pain centre at Zealand University Hospital Køge.

The patients will be tested before, halfway through, and after the programme.

DETAILED DESCRIPTION:
The number of patients with chronic non-malignant pain is high and constant. An estimated 3-5% of the population use opioids daily. These patients have a lower quality of life and a higher use of healthcare services.

This leads to enormous costs, both human and economic. Many patients lose their ability to work, not only because of the pain, but also because of their treatment.

For a long period, opioids have been prescribed for chronic pain, even though the evidence is scarce.

A rising conscience about opioid use is on the way, and now, there is a tendency to reduce, rather than increase opioids.

The reasons are many: Constipation, inability to drive, a sense of drowsiness and no relief of pain, just to name a few. Furthermore, opioids may have decreased effect over time or may even lead to higher levels of pain.

Many patients are at first reluctant to start the reduction programme. Mostly because the patients may not be aware of the effects, the drugs are having on them. Many patients value their opioid treatment as positive and necessary, in spite of the many adverse effects.

The investigators wanted to test the cognitive function of patients before, during and after opioid reduction. The results can be used to help patients understand the deleterious effects of high opioid usage, and can also be used to motivate the individual patient along the way.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age and able to provide a written consent
* Participating in the opioid reduction programme

Exclusion Criteria:

* Not able to speak and understand Danish
* Patients suffering from dementia or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain, treated with opioids and participating in the opioid reduction programme at the Multidiscipinary Pain Centre at Zealand University Hospital Køge
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Cognitive function before opioid reduction | At first visit to pain clinic (Day 1)(Individual date, inclusion is possible throughout study period)
  Cognitive function measured with the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)

SECONDARY OUTCOMES:
Cognitive function at halfway point | When opioids are reduced to half the dose (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 6 months)
  Cognitive function measured with the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Cognitive function at end of reduction | When reduction is complete (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 12 months)
  Cognitive function measured with the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
Executive function before opioid reduction | At first visit to pain clinic (Day 1)(Individual date, inclusion is possible throughout study period)
  Executive function measured by Trail making test A and B
Executive function at halfway point | When opioids are reduced to half the dose (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 6 months)
  Executive function measured by Trail making test A and B
Executive function at end of reduction | When reduction is complete (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 12 months)
  Executive function measured by Trail making test A and B
Morphine use before reduction | At first visit to pain clinic (Individual date, inclusion is possible throughout study period)
  Morphine equivalents before reduction
Morphine use after reduction | At end of reduction (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 12 months)
  Morphine equivalents after reduction
Use of other analgesics before reduction | At first visit to pain clinic (Day 1)(Individual date, inclusion is possible throughout study period)
  Use of any other analgesic
Use of other analgesics at halfway point | When opioids are reduced to half the dose (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 6 months)
  Use of any other analgesic
Use of other analgesics after reduction | At end of reduction (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 12 months)
  Use of any other analgesic
Quality of life before reduction | At first visit to pain clinic (Day 1)(Individual date, inclusion is possible throughout study period)
  Quality of life measured by SF36
Quality of life at halfway point | When opioids are reduced to half the dose (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 6 months)
  Quality of life measured by SF36
Quality of life at end of reduction | At end of reduction (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 12 months)
  Quality of life measured by SF36
Risk of anxiety and depression before reduction | At first visit to pain clinic (Day 1)(Individual date, inclusion is possible throughout study period)
  Risk of anxiety and depression measured by Hospital anxiety and depression scale
Risk of anxiety and depression at halfway point | When opioids are reduced to half the dose (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 6 months)
  Risk of anxiety and depression measured by Hospital anxiety and depression scale
Risk of anxiety and depression at end of reduction | At end of reduction (Opioid tapering is an individual process, and thus the time frame is individual, based upon morphine-reduction regimen, approximately 12 months)
  Risk of anxiety and depression measured by Hospital anxiety and depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Stine Estrup, MD, Principal Investigator — Zealand University Hospital
Locations (2):
- Denmark (2):
  - Holbæk Hospital, Holbæk
  - Zealand University Hospital, Køge

IPD SHARING:
Plan to Share IPD: No